CLINICAL TRIAL: NCT05907213
Title: Ketamine Tolerated Dose for Postpartum Depression and Pain After Cesarean Delivery (PREPARE1)
Brief Title: Ketamine Tolerated Dose for Postpartum Depression and Pain After Cesarean Delivery (PREPARE 1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grace Lim, MD, MS (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Grace Lim, MD, MS, Associate Professor, Chief Obstetric & Women's Anesthesiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: STUDY22100018; R01MH134538 (NIH)
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Pain, Postoperative; Depression, Postpartum
Keywords: Cesarean Delivery
MeSH Terms: conditions — Pain, Postoperative; Depression, Postpartum | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: MTD 3+3 design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ketamine (Ketalar) Dose Level 1 (Experimental): Ketamine (Ketalar) Dose Level 1: Loading Dose: 0.05 mg/kg/hr X 1 hour; Maintenance Dose 0.05 mg/kg/hr x 12 hours
  Interventions: Drug: Ketamine (Ketalar) Dose Level 1
- Ketamine (Ketalar) Dose Level 2 (Experimental): Ketamine (Ketalar) Dose Level 2: Loading Dose: 0.08 mg/kg/hr X 1 hour; Maintenance Dose 0.05 mg/kg/hr x 12 hours
  Interventions: Drug: Ketamine (Ketalar) Dose Level 2
- Ketamine (Ketalar) Dose Level 3 (Experimental): Ketamine (Ketalar) Dose Level 3: Loading Dose: 0.12 mg/kg/hr X 1 hour; Maintenance Dose 0.05 mg/kg/hr x 12 hours
  Interventions: Drug: Ketamine (Ketalar) Dose Level 3
- Ketamine (Ketalar) Dose Level 4 (Experimental): Ketamine (Ketalar) Dose Level 4: Loading Dose: 0.18 mg/kg/hr X 1 hour; Maintenance Dose 0.05 mg/kg/hr x 12 hours
  Interventions: Drug: Ketamine (Ketalar) Dose Level 4

INTERVENTIONS:
Drug: Ketamine (Ketalar) Dose Level 1 — Loading Dose: 0.05 mg/kg/hr X 1 hour; Maintenance Dose 0.05 mg/kg/hr x 12 hours
  Other Names: 0.05 mg/kg/1hr loading dose Ketamine
  Arms: Ketamine (Ketalar) Dose Level 1
Drug: Ketamine (Ketalar) Dose Level 2 — Loading Dose: 0.08 mg/kg/hr X 1 hour; Maintenance Dose 0.05 mg/kg/hr x 12 hours
  Other Names: 0.08 mg/kg/1hr loading dose Ketamine
  Arms: Ketamine (Ketalar) Dose Level 2
Drug: Ketamine (Ketalar) Dose Level 3 — Loading Dose: 0.12 mg/kg/hr X 1 hour; Maintenance Dose 0.05 mg/kg/hr x 12 hours
  Other Names: 0.12 mg/kg/1hr loading dose Ketamine
  Arms: Ketamine (Ketalar) Dose Level 3
Drug: Ketamine (Ketalar) Dose Level 4 — Loading Dose: 0.18 mg/kg/hr X 1 hour; Maintenance Dose 0.05 mg/kg/hr x 12 hours
  Other Names: 0.18 mg/kg/1hr loading dose Ketamine
  Arms: Ketamine (Ketalar) Dose Level 4

SUMMARY:
The purpose of this study is to identify a tolerable dose for postpartum ketamine infusion using a maximum tolerated dose (MTD) 3+3 design. A loading dose over 1 hour will be the MTD variable to be tested, as our data suggest that ketamine side effects occur with the loading dose. The investigators hypothesize that subanesthetic ketamine dose will be well tolerated and any noted side effects will be rated acceptable by postpartum women following cesarean delivery.

DETAILED DESCRIPTION:
Pain management for women having a cesarean delivery is rather limited and risks poor pain control, depressed mood, and poor recovery following the cesarean delivery. Current cesarean pain management treatments ignore the multidimensionality of pain, including the influence of mood on pain. Recent evidence suggests that ketamine may provide successful post-surgical pain management, opioid reduction, and rapid reduction of depressive symptoms. The current study aims to identify an appropriate dose of ketamine for post-cesarean pain management while minimizing potential dose-dependent side effects in women following childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* Cesarean Delivery
* American Society of Anesthesiologists Physical Status of 2 or 3
* Neuraxial anesthesia with neuraxial morphine
* Term delivery ≥37 weeks gestation
* Either planning not to breastfeed, OR receiving ketamine as part of routine clinical care

Exclusion Criteria:

* General anesthesia
* Allergy to study medications
* ASA PS 4 or higher
* Contraindications to neuraxial anesthesia
* Preterm delivery (<37 weeks gestation)
* Anticipated fetal-neonatal complex care plan
* Participating in another pain intervention trial
* Hypertensive disorder of pregnancy
* Pre-eclampsia with severe features
* Hemodynamic instability
* Medical History exclusions: ketamine or PCP (phencyclidine) abuse, schizophrenia or psychosis, liver or renal insufficiency, uncontrolled hypertension, chest pain, arrhythmia, head trauma, or intracranial hypertension, uncontrolled thyroid disease, or other contraindications to ketamine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lim, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available for public benefit and knowledge. Items for uploading will include clinical measures, patient reported outcomes, psychometric testing data, sensory testing data, and all PK data. Technical protocols and any other data collected under this project will be shared upon request to allow others to perform secondary analyses.
Supporting Information: Study Protocol, CSR
Time Frame: Beginning with 3 months and ending at 5 years following article publication.
Access Criteria: Researchers who propose a methodologically sound proposal may submit said proposals to limkg2@upmc.edu. To gain access to data, requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine (Ketalar) Dose Level 1 | Ketamine (Ketalar) Dose Level 2 | Ketamine (Ketalar) Dose Level 3 | Ketamine (Ketalar) Dose Level 4
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine (Ketalar) Dose Level 1 | Ketamine (Ketalar) Dose Level 2 | Ketamine (Ketalar) Dose Level 3 | Ketamine (Ketalar) Dose Level 4 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (3.2) | 35.3 (6.0) | 32.0 (3.6) | 33.0 (1.7) | 34.3 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 3 | 12
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 2 | 3 | 2 | 2 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 12
Estimated Gestational Age at Delivery [Count of Participants; unit: Participants]
  37-weeks | 0 | 0 | 1 | 1 | 2
  38-weeks | 0 | 1 | 0 | 0 | 1
  39-weeks | 3 | 1 | 2 | 2 | 8
  40-weeks | 0 | 1 | 0 | 0 | 1
History of Anxiety [Count of Participants; unit: Participants] | 1 | 0 | 2 | 1 | 4
History of Depression [Count of Participants; unit: Participants] | 2 | 3 | 1 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Ketamine
Description: Maximum tolerated dose of ketamine is measured by dose that fewer than 33% of patients experience a dose-limiting toxicity (DLT) defined by intolerability. Tolerability will be defined as: lack of adverse events (adverse event defined as: severe unresolved hemodynamic effect: systolic blood pressure <80 or >160, heart rate <40 or >120). Intolerability will be defined as presence of any adverse event (i.e., severe unresolved hemodynamic effect: systolic blood pressure <80 or >160, heart rate <40 or >120). Outcome measure of tolerability and intolerability will be reported as n (%). The MTD was 0.18 mg/kg/hr for one hour, followed by 0.05 mg/kg/hr for 11 hours.
Time Frame: Between 0 to 24 hours postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine (Ketalar) Dose Level 1 | Ketamine (Ketalar) Dose Level 2 | Ketamine (Ketalar) Dose Level 3 | Ketamine (Ketalar) Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants
  Tolerability of Dose | 3 | 3 | 3 | 3
  Intolerability of Dose | 0 | 0 | 0 | 0

2. Secondary Outcome: Patient Reported Acceptability of Any Reported Side Effects
Description: Number (%) of patient cohort reporting acceptability at each ketamine dose. Patient reported acceptability was recorded from a 21-question survey that reviewed seven common side effects: dizziness, lightheadedness, bad dreams, hallucinations, nausea, vomiting, and itchiness. Unacceptability is defined as patients reporting any of seven side effects as unacceptable.
Time Frame: Between 0 to 24-hours postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine (Ketalar) Dose Level 1 | Ketamine (Ketalar) Dose Level 2 | Ketamine (Ketalar) Dose Level 3 | Ketamine (Ketalar) Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants
  Acceptability of dose side effects | 3 | 2 | 3 | 3
  Unacceptability of dose side effects | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of enrollment (36+ weeks gestation) to 12-weeks postpartum for each enrolled participant.
Arm/Group | Ketamine (Ketalar) Dose Level 1 | Ketamine (Ketalar) Dose Level 2 | Ketamine (Ketalar) Dose Level 3 | Ketamine (Ketalar) Dose Level 4
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (Ketalar) Dose Level 1 (N=3) | Ketamine (Ketalar) Dose Level 2 (N=3) | Ketamine (Ketalar) Dose Level 3 (N=3) | Ketamine (Ketalar) Dose Level 4 (N=3)
Side effect: Itchiness (Social circumstances) | 3 (18) | 1 (14) | 1 (10) | 1 (4) — Patient reported itchiness
Side effect: Nausea/vomiting (Gastrointestinal disorders) | 2 (3) | 2 (6) | 2 (2) | 1 (1) — Patient reported nausea and/or vomiting
Side effect: Dizziness or lightheadedness (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) — Patient reported dizziness and/or lightheadedness
LSD Dysphoria Scale Score (Psychiatric disorders) | 0 | 0 | 2 | 0 — LSD scale is used occasionally as an indicator of dysphoria (negative mood or confusion) - patient reported score of >8.
Bad Dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT05907213/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT05907213/ICF_001.pdf